CLINICAL TRIAL: NCT01628315
Title: Assessment of Lesion Activity Analysis in the Avonex- Steroid Azathioprine (ASA) Study
Acronym: ASA
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Collaborators: Charles University, Czech Republic (Other); General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Buffalo Neuroimaging Analysis Center, Professor, University at Buffalo
Other Study IDs: ASA
Record Dates: First submitted 2012-05-01; First posted 2012-06-26 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis, Relapsing-remitting
Keywords: Multiple Sclerosis; ASA; MRI; Lesion activity
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mulitple Sclerosis: Patients with relapsing-remitting MS who had a MRI as part of their participation in the ASA study.
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — Annual MRIs as part of participation in the ASA study.

SUMMARY:
* To examine short- and long-term value of appearance of new active lesions in predicting extent of cortical and subcortical deep gray matter (SDGM) atrophy over 5 years in ASA (Avonex- Steroid-Azathioprine)study.
* To explore how accumulation of cortical and SDGM atrophy over 5 years differs with respect to the number of new active lesions or amount of disease activity, in early relapsing-remitting multiple sclerosis (RRMS) patients who did or did not develop sustained disability progression.
* To examine the relationship between development of cortical and SDGM atrophy and regional likelihood of development of new active lesions over 5 years.

DETAILED DESCRIPTION:
Historically, MS has been classified as a disease predominantly affecting the white matter (WM) of the central nervous system. However, pathological changes in gray matter (GM) are increasingly recognized as an important component of the MS disease process. Advances in MRI have enabled detection of changes in GM morphology.

The ASA study was a placebo-controlled trial that evaluated efficacy of Avonex® alone and in combination with azathioprine (AZA) or AZA and corticosteroids as initial MS therapy in 181 patients with early RRMS over 5 years. The study was conducted in the Czech Republic, and all clinical and MRI examinations were concluded at 5 years.

No study has evaluated the evolution of cortical and SDGM atrophy in relation to global or regional accumulation of active lesions and/or occurrence of relapses both from predictive short- and long-term perspective. The ASA study provides a unique opportunity to prospectively study the impact of cortical and SDGM atrophy accumulation on long-term disability progression in a defined cohort of early RRMS patients who presented with various amount of disease activity, as measured by the appearance of new active lesions and occurrence of relapses.

By assessing lesion activity in the 0-6 and 6-12 months in the ASA study we will be able to evaluate predictive value for development of cortical and SDGM atrophy in early RRMS patients over 5 years with respect to the number of new active lesions or amount of disease activity in the first year. We will also evaluate lesion development from 12-60 months in relation to development of cortical and SDGM atrophy. We will also analyze accumulation of cortical and SDGM atrophy in early RRMS patients who will or will not develop sustained disability progression, based on the number of new active lesions or amount of clinical and MRI disease activity in short- and long-term. Regional classification of new active lesions over 5 years in cortical, subcortical and fossa posterior will allow prospective examination of cortical and SDGM atrophy and appearance of the new lesions.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled into the 2-year, double-blind, placebo-controlled ASA study and entered 3 year extension study
* MRI was performed on all patients using a 1.5 T magnet

Exclusion Criteria:

* MRI images unable to be processed
* All 5 MRI time points not collected

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: * Multiple Sclerosis, relapsing-remitting
  * Enrolled into the 2-year, double-blind, placebo-controlled ASA study
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Lesion Activity | 5 years
  Assessment of lesion activity in the 0-6 and 6-12 months in the ASA study will allow the classification of patients with respect to the number of new active lesions over short-term (over 1 year) in order to examine predictive value of MRI disease activity in relation to development of long-term (5 year) cortical and SDGM atrophy.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zivadinov, MD,PhD,FAAN, Principal Investigator — Buffalo Neuroimaging Analysis Center
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States

REFERENCES:
- [Background] Horakova D, Dwyer MG, Havrdova E, Cox JL, Dolezal O, Bergsland N, Rimes B, Seidl Z, Vaneckova M, Zivadinov R. Gray matter atrophy and disability progression in patients with early relapsing-remitting multiple sclerosis: a 5-year longitudinal study. J Neurol Sci. 2009 Jul 15;282(1-2):112-9. doi: 10.1016/j.jns.2008.12.005. Epub 2009 Jan 24. PMID 19168190
- [Background] Horakova D, Cox JL, Havrdova E, Hussein S, Dolezal O, Cookfair D, Dwyer MG, Seidl Z, Bergsland N, Vaneckova M, Zivadinov R. Evolution of different MRI measures in patients with active relapsing-remitting multiple sclerosis over 2 and 5 years: a case-control study. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):407-14. doi: 10.1136/jnnp.2007.120378. Epub 2007 Jun 5. PMID 17550987
- [Background] Havrdova E, Zivadinov R, Krasensky J, Dwyer MG, Novakova I, Dolezal O, Ticha V, Dusek L, Houzvickova E, Cox JL, Bergsland N, Hussein S, Svobodnik A, Seidl Z, Vaneckova M, Horakova D. Randomized study of interferon beta-1a, low-dose azathioprine, and low-dose corticosteroids in multiple sclerosis. Mult Scler. 2009 Aug;15(8):965-76. doi: 10.1177/1352458509105229. Epub 2009 May 22. PMID 19465443
- [Background] Bergsland N, Horakova D, Dwyer MG, Dolezal O, Seidl ZK, Vaneckova M, Krasensky J, Havrdova E, Zivadinov R. Subcortical and cortical gray matter atrophy in a large sample of patients with clinically isolated syndrome and early relapsing-remitting multiple sclerosis. AJNR Am J Neuroradiol. 2012 Sep;33(8):1573-8. doi: 10.3174/ajnr.A3086. Epub 2012 Apr 12. PMID 22499842